CLINICAL TRIAL: NCT02295007
Title: Pilot Study to Assess Fever and Wheezing Events in Children After US Influenza Vaccines Using Text Messaging (2014-2015 Season)
Brief Title: Fever and Wheezing Events in Children After US Influenza Vaccines Using Text Messaging
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Columbia University (Other)
Collaborators: Centers for Disease Control and Prevention (U.S. Federal Agency); Boston Medical Center (Other)
Responsible Party: Principal Investigator, Melissa Stockwell, Assistant Professor of Pediatrics and Population and Family Health, Columbia University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: AAAO5253
Record Dates: First submitted 2014-11-17; First posted 2014-11-19 (Estimated); Last update posted 2016-05-12 (Estimated); Status verified 2016-05

CONDITIONS: Fever; Wheezing
MeSH Terms: conditions — Fever; Respiratory Sounds

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- text message (Other): all families will receive text messages to which they can respond to report symptoms
  Interventions: Behavioral: text message

INTERVENTIONS:
Behavioral: text message

SUMMARY:
Children 2-11 years of age who are given the influenza vaccine (inactivated influenza (IIV) or live attenuated influenza vaccine (LAIV)) as part of their routine care can enroll in this study if their parent has the ability to receive and send text messages. Children enrolled in this study will be observed daily for an eight-day period starting on the day of vaccine administration, and then continuing over the next 7 days, and then weekly for 42 days. On the day of enrollment and nightly for the next seven days, the parent will report via text message what their child's highest temperature is. If fever is present, they will then be prompted for additional information including other symptoms, antipyretic use and medical care sought. On day 3 as well as weekly from day 7 through day 42 post-vaccination, parents will be asked via text message about breathing problems, specifically cough, wheezing and chest tightness. They will also be asked about medications taken and care sought. The purpose of this study is to assess the feasibility of collecting this data.

ELIGIBILITY:
Inclusion Criteria:

1. are 2 through 11years of age,
2. have a visit at a study site anytime during the study period,
3. receive first dose or second dose of LAIV4 or IIV in the season,
4. the parent has a cell phone with text messaging capabilities, and
5. the parent and child > 7 years of age speaks English or Spanish at the Columbia sites or English at the Boston site.

Exclusion criteria:

1. presence of fever ≥100.4 at time of vaccination,
2. administration of any antipyretic in the 6-hour period prior to vaccination,
3. stated intent, at time of vaccination, to use prophylactic antipyretics before the development of a fever,
4. parent only speaks a language other than English or Spanish at the Columbia sites or English at the Boston site.
5. enrollee is a child >7 years of age who only speaks a language other than English or Spanish at the Columbia sites or English at the Boston site.
6. parent's inability to read and send text messages,
7. sibling already enrolled this season (OR cell phone # already used for another child)
8. chronic medical condition considered by ACIP to be a precaution or contraindication for LAIV1 (except for asthma),
9. current asthma exacerbation, or exacerbation in the last 2 weeks
10. use of oral or other systemic steroid within the last 2 weeks

Ages: 2 Years to 11 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 266 (Actual)
Dates: Start 2014-12; Primary Completion 2016-04 (Actual); Study Completion 2016-05 (Actual)

PRIMARY OUTCOMES:
feasibility reporting respiratory symptom | days 0-42 days post-vaccination
  Response rates to text messages regarding wheezing, cough or chest tightness symptoms

SECONDARY OUTCOMES:
feasibility reporting fever | days 0-7 days post-vaccination
  Response rates to text messages regarding temperature

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Stockwell, MD MPH, Principal Investigator — Columbia University; Philip LaRussa, MD, Principal Investigator — Columbia University
Locations (3):
- United States (3):
  - Centers for Disease Control and Prevention, Atlanta, Georgia
  - Boston Medical Center, Boston, Massachusetts
  - Columbia University, New York, New York

REFERENCES:
- [Derived] Stockwell MS, Marchant CD, Wodi AP, Barnett ED, Broder KR, Jakob K, Lewis P, Kattan M, Rezendes AM, Barrett A, Sharma D, Fernandez N, LaRussa P. A multi-site feasibility study to assess fever and wheezing in children after influenza vaccines using text messaging. Vaccine. 2017 Dec 15;35(50):6941-6948. doi: 10.1016/j.vaccine.2017.10.073. Epub 2017 Oct 28. PMID 29089191